CLINICAL TRIAL: NCT06934317
Title: Maximum Occlusal Bite Force of Necrotic Mature and Immature Permanent Teeth pre-and Post-treatment With the Available Treatment Modalities: Randomized Clinical Trial
Brief Title: Maximum Occlusal Bite Force of Necrotic Permanent Teeth Treated by Regenerative Technique: Randomized Clinical Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lama Awawdeh (Other)
Responsible Party: Sponsor-Investigator, Lama Awawdeh, Professor, King Abdullah University Hospital
Organization: King Abdullah University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KingAbdullahUH3
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Necrotic Pulp; Regenerative Endodontic Procedures; Bite Force
Keywords: regenerative endodontic; maximum bite force
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Induced bleeding mature and immature group (Experimental): Regeneration procedures will be conducted in two appointments, adhering to the 'Clinical Considerations for a Regenerative Procedure' proposed by the American Association of Endodontists (AAE) in 2021. All cases will receive a permanent restoration as a final restoration and a post-operative periapical radiograph
  Interventions: Diagnostic Test: measurement of maximum bite force using bite fork; Procedure: pulp revascularization by induced bleeding
- root canal treated mature group (Placebo Comparator): conventional root canal treatment in mature necrotic teeth with periapical lesion
  Interventions: Diagnostic Test: measurement of maximum bite force using bite fork; Procedure: conventional root canal treatment
- MtA apexification (Placebo Comparator): which includes the immature necrotic permanent teeth, will randomly receive either MTA apexification or revascularization
  Interventions: Diagnostic Test: measurement of maximum bite force using bite fork; Procedure: MTA apexification

INTERVENTIONS:
Diagnostic Test: measurement of maximum bite force using bite fork — using bite fork the bite force will be recorded for all teeth preoperative and post operative
Procedure: conventional root canal treatment — General principles of conventional endodontic treatment will be applied in all cases, such as the administration of an appropriate local anaesthetic and rubber dam isolation. access and cleaning and shaping using rotary files and obturation. All cases will receive a permanent restoration as a final restoration and a post-operative periapical radiograph
  Arms: root canal treated mature group
Procedure: pulp revascularization by induced bleeding — Regeneration procedures will be conducted in two appointments, adhering to the 'Clinical Considerations for a Regenerative Procedure' proposed by the American Association of Endodontists (AAE) in 2021. All cases will receive a permanent restoration as a final restoration and a post-operative periapical radiograph
  Arms: Induced bleeding mature and immature group
Procedure: MTA apexification — MTA apical plug will be randomly applied to teeth with open apex
  Arms: MtA apexification

SUMMARY:
Further investigation is warranted to ascertain whether the regaining of sensibility and nerve function in regenerated teeth leads to the re-establishment of the proprioceptive protective mechanism inherent in vital teeth.

Hence, the primary objective of this prospective randomized clinical trial is to conduct a comparative analysis of the potential effects of pulp revascularization in comparison to conventional endodontic treatments, either RCT or apexification on the Maximum occlusal bite force (MBF) in both immature and mature necrotic permanent teeth.

Methods: Upon satisfying the predetermined criteria for inclusion, a total of 184 patients will be recruited for this prospective clinical trial. The study will consist of two groups, specifically Group I: Mature teeth and Group II: Immature teeth, with a sample size of 92 participants in each group. The participants will be assigned randomly to one of the two treatment modalities per group. Group I: will undergo treatment with RCT/revascularization, while Group II will receive MTA plug/revascularization encompassing both mature (n=92) and immature teeth (n=92). MBF will be measured on the selected necrotic teeth prior to clinical intervention, this measurement will be conducted using a portable occlusal force gauge (GM10). Following the completion of therapy, MBF measurements will be repeated at 6 and 12 months to assess long-term outcomes. Subsequently, the collected data will undergo comprehensive analysis.

DETAILED DESCRIPTION:
The maximum bite force (MBF) or masticatory force results from the contact of the maxillary and mandibular teeth with the bones and muscles of the jaw [1,2,3].

Although, it is well known that the protective reflex with the jaw elevator muscle is initiated through the activation of mechanoreceptors located within the periodontal ligament [3,4,5,6]. Several studies in the literature have provided compelling evidence supporting the involvement of dental pulp in the reflex withdrawal reaction and its ability to mediate proprioceptive functions via intradental mechanoreceptors. These mechanoreceptors play a crucial role in transmitting tactile impulses through fast conducting A-delta and A-beta fibres, ultimately reaching the principal sensory nucleus of the trigeminal nerve [7-11].

Henceforth, subsequent carrying out of root canal treatment (RCT) and apexification, which are widely recognised as conventional treatment approaches for necrotic mature and immature teeth respectively, it seems that a portion of the protective mechanism and stress reduction effect is compromised due to the removal of pulpal tissue [12]. Consequently, diminished ability to control the strain exerted on dentin, along with changes in the mechanical and physical characteristics of dentin and loss of tooth structure during cavity preparation and instrumentation. Thus, the tooth becomes more susceptible to occlusal forces, thereby elevating the risk of fracture [13-15]. This has been tested by previous studies, which have demonstrated that MBF is greater in teeth that have undergone endodontic treatment than in vital contralateral teeth [8,16]. Therefore, the alternative path in which endodontics is moving is towards regenerative endodontic procedures (REPs) rather than replacing tissues with artificial alternatives.

Regenerative endodontic procedures are defined as "biologically based procedures designed to replace damaged structures, including dentin and root structures, as well as cells of the pulp-dentin complex" [17]. It capitalizes on the presence of undifferentiated mesenchymal stem cells (MSCs) within the periapical tissues. These cells gain access to the root canal after over-instrumentation of the apex [18]. Additionally, the growth factors present in the dentine play a pivotal role in directing the migration, proliferation, and differentiation of these stem cells, which possess the ability to regenerate the pulp-dentin complex.

REPs have been widely recognized as a clinically effective treatment modality, as numerous clinical studies and case reports have shown favorable outcomes in terms of root development, apical closure, periapical lesion healing, and symptoms resolution in the majority of treated mature and immature teeth [19-26].

The question arises as to the status of neural regeneration, there is a strong evidence that show that the formed pulp-like tissue after REPs has a sensory innervation, treated cases have demonstrated positive responses to sensibility tests, including cold or electric pulp test, indicating the potential reinnervation of the regenerated tissues [27, 28]. A study by Diogenes indicated that these vitality responses require targeting of the periapical neuronal terminals into coronal areas of the repaired tissue nearly 10-15 mm away from the closest nerve trunks [29]. A histological examination revealed the presence of organised nerve fibres in two teeth treated with REP [30], and another recent study demonstrated the presence of sensory fibers after REP of necrotic pulp [31].

Regaining sensitivity and nerve fibers suggested regaining the nerve function and pulp's proprioceptive defense against occlusal forces which will protect the pulp from damage and increases tooth fracture resistance [28].

Performance of revitalized teeth against occlusal loading has been studied by Finite element analysis (FEA), one study using 3D FEA that were developed from CBCT scans shows that immature teeth treated with revascularization has lower stress values and risk of fracture due to continual root development and change in root dimensions [32]. Another study concluded that following pulp revascularization, the deposition of dentin exhibits a substantial enhancement in mechanical resistance, this consequently leads to a more uniform distribution of stress during biting scenarios, as opposed to the condition observed in immature teeth [33].

Various devices have been employed to directly measure bite force in scientific studies, such as the bite fork, strain gauge transducers, foil transducers, the pressurized rubber tube, the gnathodynamometer, the pressure-sensitive sheet, and force sensing resistors. The present study aims to assess bite force using a bite fork device (GM10), which incorporates a hydraulic pressure gauge. Prior investigations have demonstrated that the aforementioned bite fork exhibits noteworthy test-retest reliability and has been validated by prior scholarly inquiries, thus establishing its suitability for facilitating endodontic clinical trials [16].

The research significance lies in the evident gap within the current body of knowledge concerning the biomechanical characteristics of teeth subjected to REPs versus conventional treatments. Furthermore, the limited available data on the capacity of regenerated pulp tissue, post-revascularization, to restore the pulp's proprioceptive defense against occlusal forces underscores the need for this investigation.

This prospective clinical trial involves measurements of MBF in necrotic mature and immature teeth undergoing either RCT or apexification, as well as revascularization. By doing so, it aims to shed light on the role of pulp revascularization in modulating occlusal loads in both mature and immature teeth. This examination of how regenerated pulp tissues may influence bite force values promises to provide valuable insights into this crucial aspect. Moreover, this methodology also serves to validate findings from previous studies exploring the impact of pulp on regulating bite force measurements

ELIGIBILITY:
Inclusion Criteria:

* Healthy (ASA Grade 1 & 2 status). Compliant patient/parent. Mature and immature teeth diagnosed with necrotic pulp. Pulp space is not needed for post and core restoration for cases treated by revascularization.

Patients are not allergic to the medications necessary to complete the procedure.

The presence of opposing teeth for the included necrotic teeth. No medication (steroids) at the time of investigation, and the patient should not have taken analgesics 6 hours ago.

Exclusion Criteria:

* Medically compromised patient. Patient with generalized chronic periodontitis. Patient with TMD. Current orthodontic treatment. Teeth with sensitivity to percussion. Teeth with previous root canal treatment. Periodontal pocket more than 3mm. Teeth with vertical fractures. Teeth with large restorations, either direct or indirect restoration Teeth with large carious lesions. Non-restorable teeth.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
clinical signs and symptoms | in 3, 6 and 12 months intervals
  absence of pain, tenderness, and evidence of radiographic healing

SECONDARY OUTCOMES:
assesment of pulp vitality | in 6 and 12 months intervals
  using positive respone to cold test and electirc pulp tester

OTHER OUTCOMES:
maximum bite force | in 6 and 12 months intervals
  bite force will be measured using a bite fork pre-operatively and post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Dental Clinic Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided